CLINICAL TRIAL: NCT00988897
Title: A Phase II Study of Modified FOLFOX-6 Chemotherapy as First-line Treatment of Metastatic Colorectal Cancer in Patients Who Have Received Oxaliplatin-based Adjuvant Chemotherapy
Brief Title: Colorectal Cancer RECHALLENGE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_03943
Record Dates: First submitted 2009-09-28; First posted 2009-10-02 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Bevacizumab

ARMS (1):
- 1 (Experimental): Patients will receive modified FOLFOX-6 regimen:
  * oxaliplatin 85mg/m2, day 1 (given as a 2-hour infusion)
  * LV 400mg/m2, day 1 (given as a 2-hour infusion simultaneous to oxaliplatin)
  * 5-FU given as a bolus IV 400mg/m2 dose on day 1 followed by 2400mg/m2 continuous infusion over 46 hours (day 1 and 2)
  A cycle is defined as 2 weeks. Patients will receive cycles of modified FOLFOX-6 regimen every 2 weeks up to a maximum of 8 cycles. Use of bevacizumab is at the discretion of the treating physician.
  Interventions: Drug: OXALIPLATIN (SR96669); Drug: 5-FLUOROURACIL (5-FU); Drug: LEUCOVORIN (LV); Drug: BEVACIZUMAB

INTERVENTIONS:
Drug: OXALIPLATIN (SR96669) — Pharmaceutical form: Lyophilized powder for injection (50mg/vial or 100mg/vial) or aqueous solution (50mg/10mL or 100mg/20mL) Route of administration: IV
Drug: 5-FLUOROURACIL (5-FU) — Pharmaceutical form: vials of 5g/100mL (50mg/mL) Route of administration: IV
Drug: LEUCOVORIN (LV) — Pharmaceutical form: vials of 50mg/5mL or 500mg/50mL (10mg/mL) Route of administration: IV
Drug: BEVACIZUMAB — Pharmaceutical form: vials of 100mg/4mL or 400mg/16mL (25mg/mL) Route of administration: IV

SUMMARY:
Primary Objective:

* To demonstrate that re-challenge with an oxaliplatin based regimen (modified FOLFOX-6) will provide a clinical disease control rate (DCR) of at least 20% at the end of the chemotherapy.

Secondary Objective:

* To evaluate other measures of tumour's responses and safety.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven adenocarcinoma of colon or rectum
* Measurable metastatic disease, either inoperable, or residual after surgical procedure
* No prior chemotherapy for metastatic disease
* For colon cancer: prior adjuvant chemotherapy with oxaliplatin that ended at least 12 months prior to enrollment.
* For rectal cancer: at least 12 months since prior use of oxaliplatin in neoadjuvant or adjuvant chemotherapy
* Adequate liver and kidney function:

  * Total bilirubin inferior to 1.5 ULN
  * Serum Creatinine inferior to 150 umol/L
  * Creatinine clearance (ClCr) > 30 mL/min
  * ALT / AST inferior to 3 ULN
* Adequate hematological function

  * Neutrophils > or equal 1.5 x 109/L
  * Platelets > or equal 100 x 109/L

Exclusion criteria:

* Metastatic disease presenting without prior adjuvant chemotherapy
* Metastatic disease presenting after non-oxaliplatin-containing adjuvant chemotherapy
* Peripheral sensory or motor neuropathy > grade 1
* Eastern Cooperative Oncology Group (ECOG) Performance status > 2
* Other active malignancy
* History of known allergy to oxaliplatin or other platinum compounds, to 5-FU, to Leucovorin or to any ingredients in the formulations or the containers
* Patients who are pregnant, or breast-feeding
* Patients with severe renal impairment (ClCr < 30 mL/min)
* Pernicious anemia or other megaloblastic anemia with Vitamin B12 deficiency
* Patients with reproductive potential not implementing accepted and effective method of contraception (the definition of effective method of contraception will be based on the investigators' judgment)
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening
* For patient who will receive Bevacizumab: Bevacizumab is contraindicated in patients with know hypersensitivity to any components of the product and to Chinese hamster ovary cell product or other recombinant human or humanized antibodies
* Presence of any symptoms suggesting brain metastasis

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint for the first thirteen patients according to the Simons Design: Clinical DCR (Disease Control Rate) at the end of stage I, based on Response Evaluation Criteria on Solid Tumors (RECIST) criteria. | At the end of 8 cycles or end of treatment which occurs first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | evaluated at 10 weeks, 16 weeks and 40 weeks
Duration of response | evaluated at 10 weeks, 16 weeks and 40 weeks
Adverse events | At each visit, i.e. every two weeks
Overall response rate of stage I and II | evaluated at week 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada